CLINICAL TRIAL: NCT05808205
Title: An Open, Non-comparative, Single-centre Post Marketing Clinical Follow-up (PMCF) Investigation to Evaluate Performance and Safety of the ALIAXIN Fillers Used as Intended
Brief Title: An Open, Non-comparative, Single-centre Post Marketing Clinical Followup (PMCF) Investigation to Evaluate Performance and Safety of the ALIAXIN Fillers Used as Intended
Status: Recruiting | Type: Observational
Sponsor: Rose Pharma SA (Industry)
Responsible Party: Sponsor
Other Study IDs: RP-ALX-01_2019
Record Dates: First submitted 2023-02-28; First posted 2023-04-11 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Esthetics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Open Non-comparative: In this study, it is planned to include about 70 patients each year, assuming two treatments per patient. Due to the post-market nature of the study, this sample size is not based on a formal statistical sample size calculation, but the size is considered appropriate for the study purposes and considering the enrollment rate estimated at the center.
  Interventions: Device: • ALIAXIN EV: Essential Volume • ALIAXIN FL: Lips • ALIAXIN SR: Shape & Restore • ALIAXIN GP: Global Performance • ALIAXIN LV: Lips Volume

INTERVENTIONS:
Device: • ALIAXIN EV: Essential Volume • ALIAXIN FL: Lips • ALIAXIN SR: Shape & Restore • ALIAXIN GP: Global Performance • ALIAXIN LV: Lips Volume — According the investigator judgment and IP' Instruction For Use (IFU), each subject can be treated in one or more of following face area:
  * Temporal / frontal area
  * Orbital / Malar area
  * Perioral area
  * Lips.

SUMMARY:
This is an open, non-comparative, Single-centre Post Marketing Clinical Followup (PMCF) study aimed to enrol patients with medium and deep facial sagging, facial volume defects and/or lips volume and contours defects. The investigation will be useful to collect Investigational Product' real world safety /performance evidences in normal clinical practice. Each subject, after signing the Informed Consent, will enter into a 1-week screening phase during which the baseline tests will be conducted. At baseline visit (Visit 0), as per clinical practice, the subject can be treated with one or more of the below ALIAXIN products, depending on investigator clinical evaluation and decision:

* ALIAXIN EV: Essential Volume
* ALIAXIN FL: Lips
* ALIAXIN SR: Shape & Restore
* ALIAXIN GP: Global Performance
* ALIAXIN LV: Lips Volume According the investigator judgment and IP' Instruction For Use (IFU), each subject can be treated in one or more of following face area:
* Temporal / frontal area
* Orbital / Malar area
* Perioral area
* Lips. For the pre- and post-treatment clinical evaluations, a LifeViz® Mini 3D camera (QuantifiCare) will be used for face-images capture. A LifeViz® Micro 3D camera (QuantifiCare) will be used for adjuvant images capture, only in specific conditions (e.g. nasolabial folds and marionette lines) and according to the Principal Investigator judgment, to facilitate the clinical evaluation. As per clinical practice, the treatment can be repeated at touch up visit (Visit 1), after 15 days from Visit 0, according the investigator clinical evaluation and decision, to maintain/refine the obtained results. Moreover, after 6 months from Visit 0, as per clinical practice, a visit ( Visit 2, End of Study Visit) will be performed to collect and evaluate the safety and performance of treatment(s) performed. Considering the normal clinical practice, after Visit 2, according the investigator judgment and after a new Informed Consent Form signature, the subject can be enrolled in a new screening phase as per clinical study design. The re-enrolled subject should meet all inclusion and none exclusion criteria. In the new CRF will be reported the previous subject's identification number.

DETAILED DESCRIPTION:
Aesthetic Dermatology (AD) is a rapidly developing part of dermatology in science and clinical practice.

The focus, however, needs to be patient-centered and the work scientific to avoid the ethical dilemma.

The growing patient population and appeal for rapid results have served as an impetus that transformed the use of soft tissue fillers. While clinicians established innovative ways to address multidimensional deficiencies of the face, manufacturers developed new formulations to address the tasks faced by clinicians. With these advancements, it is essential that facial plastic surgeons are adept at cosmetic applications of soft tissue fillers to provide quality care and optimize patient outcomes.

Today, there are a variety of injectable soft tissue fillers available for clinical use with over 160 products belonging to > 50 companies on the market. Factors such as defect type and location, preferred durationof effect, and clinician expertise with specific agents determine the most approp riate choice of agent. These fillers can be categorized into resorbable (biodegradeable), nonresorbable (permanent), and viable autologous fat. Resorbable fillers include hyaluronic acid (HA), collagen, calcium hydroxylapatite, and poly-L-lactic acid with HA-based fillers being the most common injectable agents used today. Common permanent fillers include polymethylmethacrylate (PMMA) microspheres, hydrogel polymers, and silicone injections. Because most patients are satisfied with temporary filler use, the decision to pursue permanent fillers must be considered carefully.

Hyaluronic acid (HA) is a naturally occurring polysaccharide frequently used as a functional ingredient in subcutaneous antiaging treatments, such as dermal fillers, which use the polymer's unique viscoelastic properties. The major challenge lies in the reasoned choice of the product to be used depending on the anatomical area to be corrected. Indeed, each region of the face is subjected to specific mechanical constraints, which the authors take into account when selecting HA.

Hyaluronic acid can be defined by viscoelasticity and cohesiveness, which will determine the resistance to deformation during mechanical stresses.

The clinical persistence and characteristics of HA-based dermal fillers may be influenced by their physical properties. Increasing both the molecular weight and degree of cross-linking of the polymer is a proven strategy for improving mechanical strength and extending degradation times.

"ALIAXIN" is a HA-based dermal filler. It is available in five different formulations, with specific and differentiated visco-elastic properties: ALIAXIN EV (Essential Volume), ALIAXIN FL (Lips), ALIAXIN SR (Shape & Restore), ALIAXIN GP (Global Performance), ALIAXIN LV (Lips Volume). Their different behaviours, studied to treat different facial area, are deriving from the combined use of different molecular weight hyaluronic acids and their crosslinking degree.

The formulations offered by the "ALIAXIN" line are based on the concept of Hydrolift® Action: the innovative approach that aims to counteract the reduction of hyaluronic acid in the skin, restoring hydration, elasticity and skin tone.

"ALIAXIN" has been on the market for many years and in literature are available several safety and performance clinical data, collected by controlled studies, in which authors tested "ALIAXIN" or other similar HA-based dermal fillers according the intend of use.

The aim of this open, non-comparative, Single-centre Post Marketing Clinical Follow-up (PMCF) is to collect "ALIAXIN" real world safety and performance evidences in normal clinical practice, in the treatment of patients with medium and deep facial sagging, facial volume defects and/or lips volume and contours defects.

This is a Post-market clinical follow-up Medical Device study

The study objective are the following:

Primary

• To evaluate the re-volumizing performance of the filler ALIAXIN (EV, FL, SR, GP and LV) used as Intended in patients with facial volume defects.

Secondary

* To evaluate the corrective performance of the filler ALIAXIN (EV, FL, SR, GP and LV) used as Intended in patients with medium and deep facial sagging;
* To evaluate the safety, tolerability and patient satisfaction of the filler ALIAXIN (EV, FL, SR, GP and LV).

Methodology: This is an open, non-comparative, Single-centre Post Marketing Clinical Follow-up (PMCF) study aimed to enrol patients with medium and deep facial sagging, facial volume defects and/or lips volume and contours defects. The investigation will be useful to collect Investigational Product' real world safety /performance evidences in normal clinical practice.

Each subject, after signing the Informed Consent, will enter into a 1-week screening phase during which the baseline tests will be conducted.

At baseline visit (Visit 0), as per clinical practice, the subject can be treated with one or more of the below ALIAXIN products, depending on investigator clinical evaluation and decision:

* ALIAXIN EV: Essential Volume
* ALIAXIN FL: Lips
* ALIAXIN SR: Shape & Restore
* ALIAXIN GP: Global Performance
* ALIAXIN LV: Lips Volume

According the investigator judgment and IP' Instruction For Use (IFU), each subject can be treated in one or more of following face area:

* Temporal / frontal area
* Orbital / Malar area
* Perioral area
* Lips.

For the pre- and post-treatment clinical evaluations, a LifeViz® Mini 3D camera (QuantifiCare) will be used for face-images capture.

A LifeViz® Micro 3D camera (QuantifiCare) will be used for adjuvant images capture, only in specific conditions (e.g. nasolabial folds and marionette lines) and according to the Principal Investigator judgment, to facilitate the clinical evaluation.

As per clinical practice, the treatment can be repeated at touch up visit (Visit 1), after 15 days from Visit 0, according the investigator clinical evaluation and decision, to maintain/refine the obtained results.

Moreover, after 6 months from Visit 0, as per clinical practice, a visit ( Visit 2, End of Study Visit) will be performed to collect and evaluate the safety and performance of treatment(s) performed.

Considering the normal clinical practice, after Visit 2, according the investigator judgment and after a new Informed Consent Form signature, the subject can be enrolled in a new screening phase as per clinical study design. The re-enrolled subject should meet all inclusion and none exclusion criteria.

In the new CRF will be reported the previous subject's identification number.

Number of subjects (planned and analysed):

Planned: In this study, it is planned to include about 70 patients each year, assuming two treatments per patient. Due to the post-market nature of the study, this sample size is not based on a formal statistical sample size calculation, but the size is considered appropriate for the study purposes and considering the enrollment rate estimated at the center.

To ensure the evaluation of all defined areas, for each 6 months follow-up period, it is intended that the investigational site will perform a minimum of 5 evaluations for every identified facial area (i.e., Temporal / frontal area, Orbital / Malar area, Perioral area, Lips). Considering that each subject can be treated at the same time in one or more facial area, to reach the 5 evaluations per area, the number of subjects to enrol may vary in every follow-up period.

Sample size justification: Considering a study duration of 5 years, minimum 200 treatments will be evaluated. In this study, it is planned to include about 70 patients each year, assuming two treatments per patient. Due to the post-market/observational nature of the study, this sample size is not based on a formal statistical sample size calculation, but the size is considered appropriate for the study purposes and considering the enrollment rate estimated at the center.

To ensure the evaluation of all defined areas, for each 6 months follow-up period, it is intended that the investigational site will perform a minimum of 5 evaluations for every identified facial area (i.e., Temporal / frontal area, Orbital / Malar area, Perioral area, Lips). Considering that each subject can be treated at the same time in one or more facial area, to reach the 5 evaluations per area, the number of subjects to enroll may vary in every follow-up period.

Treatment duration: As per clinical practice, after baseline injection, the treatment can be repeated only at touch up visit (15 days later) according the investigator clinical evaluation and decision. After 6 months, at follow-up visit (End of Study), will be performed the last safety and efficacy evaluation.

Safety Set: this set included all enrolled patients who took at least one does of study medication.

Full Analysis Set (FAS): this set included all enrolled patients who took at least one dose of study medication, and with a baseline and at least one post-baseline performance assessment.

Investigational Product:

* ALIAXIN EV: Essential Volume
* ALIAXIN FL: Lips
* ALIAXIN SR: Shape & Restore
* ALIAXIN GP: Global Performance
* ALIAXIN LV: Lips Volume

They have the same formulation, differentiating only for viscosity in order to better act on any given district.

Dose/dosage: ALIAXIN fillers are available in a 2ml package with inside 2 sealed blisters, each containing 1 sterile pre-filled mono-use syringe of 1 ml.

Each IP contain 25mg/ml of Hyaluronic Acid (HA) as their key functional component as described below:

* ALIAXIN EV, FL, GP and LV: HA cross-linked 25mg/ml
* ALIAXIN SR: HA cross-linked 22.5mg/ml and HA natural 2.5 mg/ml

The volumetric grading printed on the syringe has an indicative value: it is left to the doctor's discretion to choose the dosage to be used for each individual case.

Administration:

Injection in the medium/deep dermis/ superficial subcutis in accordance to the indication for use.

The first administration will be performed at baseline. As clinical practice and according the medical judgment, one or more ALIAXIN filler type (i.e. EV, FL, SR, GP and LV) can be used for each enrolled subject. Moreover, one or more face area (Temporal / frontal area, Orbital / Malar area, Perioral area, Lips) can be treated at baseline Visit.

According the normal clinical practices and investigator decision, for the maintenance/refinement of obtained results it will be possible to repeat the treatment only at touch up visit (15 days after baseline treatment). The treatment should be repeated according various factors, regarding both the physiology of the patients (type of skin, individual metabolism, anatomy, age) and their lifestyle. Another element to consider is relative to the implant techniques used in the normal clinical practices.

Criteria for evaluation:

Primary efficacy endpoint:

To evaluate the re-volumizing performance of the filler ALIAXIN (EV, FL, SR, GP and LV) used as Intended in patients with facial volume defects, by treated areas calculating the volume variation (expressed as cm3) during all study duration compared to baseline volume. A 3D camera will be used to take subject' face images at all planned visits.

Secondary efficacy endpoints

* To evaluate the corrective performance of the ALIAXIN fillers (EV, FL, SR, GP and LV) used as Intended in patients with medium and deep facial sagging, performing treated area evaluation by GAIS scale during all study duration.
* To evaluate the re-volumizing performance of each Filler ALIAXIN (EV, FL, SR, GP and LV) calculating the volume variation (expressed as cm3) during all study duration compared to baseline volume. A 3D camera will be used to take subject' face images at all planned visits.
* To evaluate the tolerability and patient satisfaction of the filler ALIAXIN (EV, FL, SR, GP and LV) using a 5 Likert Scale during all study duration.

Safety:

Safety will be monitored through vital signs, facial examination and adverse events including assessment of relationship to the IP.

Time-points for efficacy and safety: Baseline (V0) and all follow up visits performed, including visits during which administration of the product was repeated.

Interim efficacy and safety analysis: Every year an interim analysis will be completed on primary and secondary endpoints to periodically evaluate the performance and safety of the ALIAXIN fillers used as Intended.

Statistical methods: Considering a study duration of 5 years, minimum 200 treatments will be evaluated.

In general, all the variables will be descriptively analyzed by treated area groups and visit (mean, median, standard deviation, minimum and maximum for continuous variables after normality check of distribution with Kolmogorov-Smirnov test, frequency distribution for categorical variables). All the analysis will be detailed in the Statistical Analysis Plan (SAP) which will be finalized in Version 1.0 before the Data Base Lock (DBL). Confidence Intervals (CI) at 95% level will be provided.

In details, the safety data will include (at least) physical examinations, vital signs and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed consent form (ICF) signed;
* M & F Aged ≥ 18 years at the time of the signature of ICF;
* Patients with medium and deep facial sagging, facial volume defects and/or lips volume and contours defects (nasolabial folds, wrinkles around the mouth facial and acne scars, glabellar wrinkles, wrinkles on the forehead, areas of the face which require enrichment of the facial tissue - cheeks, chin, cheekbones, lips - with temporary volumetric increase through growth of the soft tissues).
* Willing to follow all study procedures, including attending all site visits, tests and examinations;
* Willing to follow indications to not be exposed to make-up, excessive heat (sun, UV tanning sessions or laser) or intense cold after the treatment and until the complete absorption of swelling and reddening.

Exclusion Criteria:

* Other - different - clinical conditions of skin layers;
* Sagging and volume defects in other parts of the body different from face;
* Infective or inflammatory processes near the area of intervention;
* Presence of tendon, bone or muscular implants near the area of intervention;
* Ongoing cutaneous allergies;
* Serious and Chronical pathological skin conditions (i.e. rosacea, psoriasis, vitiligo) including diagnosticated cancer with/without ongoing antitumor therapy;
* Known hypersensitivity to cheloids;
* Allergy to device components;
* Immune system illnesses;
* Diabetes mellitus or uncontrolled systemic diseases;
* Problems with coagulation or anti-coagulating therapies in progress;
* Current treatment with substances which act on blood fluidity (eg. Aspirin, NSAID, Vitamin E);
* History of permanent filler treatment;
* Known drug and/or alcohol abuse;
* Mental incapacity that precludes adequate understanding or cooperation;
* Participation in another investigational study;
* Pregnancy Status (as per ALIAXIN products leaflet).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, it is planned to include about 70 patients each year, assuming two treatments per patient. Due to the post-market nature of the study, this sample size is not based on a formal statistical sample size calculation, but the size is considered appropriate for the study purposes and considering the enrollment rate estimated at the center. To ensure the evaluation of all defined areas, for each 6 months follow-up period, it is intended that the investigational site will perform a minimum of 5 evaluations for every identified facial area (i.e., Temporal / frontal area, Orbital / Malar area, Perioral area, Lips). Considering that each subject can be treated at the same time in one or more facial area, to reach the 5 evaluations per area, the number of subjects to enrol may vary in every follow-up period.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the re-volumizing performance of the filler ALIAXIN during all study duration compared to baseline volume. Change will be assessed. | V-1(Week -1 Screening visit), V0 (Baseline visit day 0, IP administration). V-1 and V0 may coincide. V1 (15 days from V0) and V2 (6 months from V0). Change will be assessed.
  To evaluate the re-volumizing performance of the filler ALIAXIN (Essential Volume (EV), Lips (FL), Shape & Restore (SR), Global Performance (GP) and Lips Volume (LV)) used as Intended in patients with facial volume defects, by treated areas calculating the volume variation (expressed as cm3) during all study duration compared to baseline volume. A 3D camera will be used to take subject' face images at all planned visits.

SECONDARY OUTCOMES:
To evaluate the corrective performance of the ALIAXIN fillers during all study duration by Global Aesthetic Improvement Scale (GAIS). | V0 (Baseline visit day 0, IP administration) V1 (15 days from V0) and V2 (6 months from V0).
  To evaluate the corrective performance of the ALIAXIN fillers (Essential Volume (EV), Lips (FL), Shape & Restore (SR), Global Performance (GP) and Lips Volume (LV)) used as Intended in patients with medium and deep facial sagging, performing treated area evaluation by Global Aesthetic Improvement Scale (GAIS) during all study duration. The GAIS is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, as judged by the investigator. The rating categories were "worse," "no change," "improved," "much improved," and "very much improved."
To evaluate the re-volumizing performance of each Filler ALIAXIN during all study duration compared to baseline volume. Change will be assessed. | V-1(Week -1 Screening visit), V0 (Baseline visit day 0, IP administration). V-1 and V0 may coincide. V1 (15 days from V0) and V2 (6 months from V0). Change will be assessed.
  To evaluate the re-volumizing performance of each Filler ALIAXIN (EV, FL, SR, GP and LV) calculating the volume variation (expressed as cm3) during all study duration compared to baseline volume. A 3D camera will be used to take subject' face images at all planned visits.
To evaluate the tolerability and patient satisfaction of the filler ALIAXIN during all study duration. | V0 (Baseline visit day 0, IP administration) V1 (15 days from V0) and V2 (6 months from V0).
  To evaluate the tolerability and patient satisfaction of the filler ALIAXIN (EV, FL, SR, GP and LV) using a 5 Likert Scale during all study duration (the Likert scale is a five point scale that is used to allow an individual to express how much they agree or disagree with a particular statement).

OTHER OUTCOMES:
Safety will be monitored through vital signs by Blood Pressure | V-1(Week -1 Screening visit), V0 (Baseline visit day 0, IP administration). V-1 and V0 may coincide. V1 (15 days from V0) and V2 (6 months from V0)
  Safety will be monitored through vital signs by Blood Pressure (systolic and diastolic pressures) (mmHg)
Safety will be monitored through vital signs by Heart Rate | V-1(Week -1 Screening visit), V0 (Baseline visit day 0, IP administration). V-1 and V0 may coincide. V1 (15 days from V0) and V2 (6 months from V0)
  Safety will be monitored through vital signs by Heart Rate (beats/min).
Safety will be monitored through facial examination. PI will observe the presence of erythema and hematomas | V-1(Week -1 Screening visit), V0 (Baseline visit day 0, IP administration). V-1 and V0 may coincide. V1 (15 days from V0) and V2 (6 months from V0)
  Safety will be monitored through facial examination (presence of erythema and hematomas)
Safety will be monitored through the evaluation of the adverse events. | V-1(Week -1 Screening visit), V0 (Baseline visit day 0, IP administration). V-1 and V0 may coincide. V1 (15 days from V0) and V2 (6 months from V0)
  The event, date of onset, severity, duration, and relationship to the device will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Capitanio - Istituto Auxologico Italiano IRCCS Milano, Milan, Italy